CLINICAL TRIAL: NCT01683942
Title: A New Reproducible Method of Measuring C/D Ratio of Digital Stereo Images of Optic Disc
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NesherMimouni
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Developing Novel Technique of Measuring C/D Ratio From Digital Stereo Optic Disc Images; Intraobserver Reproducibility of C/D Measurements; Interobserver Variability of C/D Measurements
Keywords: cup disc ratio measurement; digital stereo optic disc images

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Development of a novel computer software that will assist in measuring the cup/disc ratio in digital stereo optic disc images.

ELIGIBILITY:
Inclusion Criteria:

Patients who attended the Glaucoma service Patients with at least one pair of documented digital stereo optic disc images Satisfactory Quality of image allowing Cup Disc Ratio Evaluation

Exclusion Criteria:

Unsatisfactory Quality of image allowing Cup Disc Ratio Evaluation Novel software technique unable to process or analyze the image

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 consecutive digitalized optic disc photos of 250 patients attending the Glaucoma Service between 1996-2012 will be extracted from a database of optic disc photos at the Glaucoma Service of the Ophthalmology Department, Meir Medical Center, Kfar Saba, Israel.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-08